CLINICAL TRIAL: NCT05433155
Title: Nasotracheal Intubation With Videolaryngoscopy Versus Direct Laryngoscopy in Infants (NasoVISI) Trial
Brief Title: Nasotracheal Intubation With VL vs DL in Infants Trial
Acronym: NasoVISI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: Children's Hospital Colorado (Other); Seattle Children's Hospital (Other); Baylor College of Medicine (Other); Children's Medical Center Dallas (Other); Dell Children's Medical Center of Central Texas (Other); Children's National Research Institute (Other); Vanderbilt University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 22-019921
Record Dates: First submitted 2022-06-21; First posted 2022-06-27 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Intubation Complication; Intubation; Difficult or Failed; Hypoxia; Hypoxemia; Anesthesia Intubation Complication; Pediatric HD
Keywords: Laryngoscope; Video Laryngoscope; Direct Laryngoscope; Nasotracheal Intubation; First attempt success; Intubation complications; Intubation technical difficulties; Randomization; Multi-center
MeSH Terms: conditions — Hypoxia

STUDY DESIGN:
Intervention Model Description: Prospective, randomized, multi-center parallel group trial
Who Masked: Participant
Masking Description: Blinding of the device for clinicians and study staff is not feasible in this study. Participants will be blinded. The statisticians will be blinded at the time of generating the randomization schedule and remain blinded at the time of analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Videolaryngoscopy (Active Comparator): Nasotracheal intubation performed with the Storz C-Mac Video Laryngoscope
  Interventions: Device: Nasotracheal intubation
- Direct Laryngoscopy (Active Comparator): Nasotracheal Intubation performed with the standard clinical direct blades
  Interventions: Device: Nasotracheal intubation

INTERVENTIONS:
Device: Nasotracheal intubation — Nontracheal intubation using clinical standard videolaryngoscopy or direct laryngoscopy

SUMMARY:
Nasotracheal Intubation with Videolaryngoscopy versus Direct Laryngoscopy in Infants (NasoVISI) Trial is a prospective randomized multicenter study. The study will be conducted at 8 centers in the United States. It is expected that approximately 700 subjects enrolled to product 670 evaluable subjects.The randomization is 1:1 naso tracheal intubation with the Storz C-Mac Video Videolaryngoscopy (VL) or the Standard Direct Laryngoscope (DL). The primary objective is to compare the nasotracheal intubation (NTI) first attempt success rate using VL vs. DL in infants 0-365 days of age presenting for cardiothoracic surgery and cardiac catheterizations.

DETAILED DESCRIPTION:
The primary objectives of the study are to compare the nasotracheal intubation (NTI) first attempt success rate using VL vs. DL in infants 0-365 days of age presenting for cardiothoracic surgery and cardiac catheterizations.

Secondary Objectives include the number of attempts for successful intubation; Incidence of failed NTI (conversion to oral intubation); Incidence of failure to intubate with assigned device; Incidence of complications over all attempts including non-severe and severe complications; Incidence of 1st-attempt complications; Need for cricoid pressure or external laryngeal manipulation, need for adjunct- (Magill forceps), rescue of one technique of the other, Percent of glottic opening (POGO) score less than 100%, intubation sequence exceeding 60 seconds and interaction analysis of weight group (i.e. ≤ median weight & > median weight (kg)), and by clinicians' experience with cardiac anesthesiology (i.e. Permanent full time team members & rotating team members) on the association between treatment and outcomes

Study Design: this is a prospective, randomized, multi-center parallel group trial

Setting/Participants: This will be a multi-center study. The target population will be infants 0-365 days of age scheduled for elective cardiothoracic surgery or cardiac catheterization requiring general anesthesia with NTI.

Study Interventions and Measures: The study intervention will be a 1:1 randomization to perform tracheal intubation with the Storz C-Mac Video Videolaryngoscopy (VL) or the Standard Direct Laryngoscope (DL).

Main study outcome measures are as follows:

* The first intubation attempt success rate with each device
* The number of attempts for successful intubation with each device
* Complications associated with intubation

ELIGIBILITY:
Inclusion Criteria:

* Males or females age 0 -365 days
* Scheduled for elective cardiothoracic surgery or cardiac catheterization procedures lasting longer than 30 minutes under general anesthesia where nasotracheal intubation will be performed by an anesthesiology clinician
* Plan to use a neuromuscular blocking drug prior to intubation as standard of care
* Parental/guardian permission (informed consent)

For clinician participants:

- Anesthesia attending, anesthesia fellows, anesthesia resident, Anesthesia Assistant (AA) or CRNA

Exclusion Criteria:

* Less than 36 weeks gestation
* Less than 2 kg
* History of difficult intubation
* History of abnormal airway
* Predictive of difficult intubation upon physical examination
* Preoperative endotracheal tube or tracheostomy
* Emergency cases

Ages: 1 Day to 365 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 680 (Actual)
Dates: Start 2022-06-06 (Actual); Primary Completion 2025-02-25 (Actual); Study Completion 2025-02-25 (Actual)

PRIMARY OUTCOMES:
VL first attempt success rate | 24 hours
  Direct observation of intubation in the OR and medical record review

SECONDARY OUTCOMES:
Number of attempts for successful intubation | 24 hours
  Direct observation of intubation in the OR and medical record review
Incidence of failed NTI (conversion to oral intubation) | 24 hours
  Direct observation of intubation in the OR and medical record review
Incidence of failure to intubate with assigned device | 24 hours
  Direct observation of intubation in the OR and medical record review
Incidence of complications over all attempts including non-severe and severe complications | 24 hours
  Direct observation of intubation in the OR and medical record review
Incidence of 1st-attempt complications | 24 hours
  Direct observation of intubation in the OR and medical record review
Incidence of additional techniques | 24 hours
  Direct observation of intubation in the OR and medical record review
Interaction analysis of weight group and by clinicians' experience with cardiac anesthesiology on the association between treatment and outcomes | 24 hours
  Direct observation of intubation in the OR and medical record review

CONTACTS AND LOCATIONS:
Overall Officials: Annery Garcia-Marcinikiewicz, MD, Principal Investigator — The Children Hospital of Philadelphia
Locations (8):
- United States (8):
  - Children's Hospital Colorado, Aurora, Colorado
  - Children's National Medical Center, Washington D.C., District of Columbia
  - The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - University of Texas at Austin Dell Children's Medical Center, Austin, Texas
  - Children's Medical Center Dallas, Dallas, Texas
  - Texas Children's Hospital, Houston, Texas
  - Seattle Children's Hospital, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fiadjoe JE, Nishisaki A, Jagannathan N, Hunyady AI, Greenberg RS, Reynolds PI, Matuszczak ME, Rehman MA, Polaner DM, Szmuk P, Nadkarni VM, McGowan FX Jr, Litman RS, Kovatsis PG. Airway management complications in children with difficult tracheal intubation from the Pediatric Difficult Intubation (PeDI) registry: a prospective cohort analysis. Lancet Respir Med. 2016 Jan;4(1):37-48. doi: 10.1016/S2213-2600(15)00508-1. Epub 2015 Dec 17. PMID 26705976
- [Background] Garcia-Marcinkiewicz AG, Kovatsis PG, Hunyady AI, Olomu PN, Zhang B, Sathyamoorthy M, Gonzalez A, Kanmanthreddy S, Galvez JA, Franz AM, Peyton J, Park R, Kiss EE, Sommerfield D, Griffis H, Nishisaki A, von Ungern-Sternberg BS, Nadkarni VM, McGowan FX Jr, Fiadjoe JE; PeDI Collaborative investigators. First-attempt success rate of video laryngoscopy in small infants (VISI): a multicentre, randomised controlled trial. Lancet. 2020 Dec 12;396(10266):1905-1913. doi: 10.1016/S0140-6736(20)32532-0. PMID 33308472
- [Background] Greene NH, Jooste EH, Thibault DP, Wallace AS, Wang A, Vener DF, Matsouaka RA, Jacobs ML, Jacobs JP, Hill KD, Ames WA. A Study of Practice Behavior for Endotracheal Intubation Site for Children With Congenital Heart Disease Undergoing Surgery: Impact of Endotracheal Intubation Site on Perioperative Outcomes-An Analysis of the Society of Thoracic Surgeons Congenital Cardiac Anesthesia Society Database. Anesth Analg. 2019 Oct;129(4):1061-1068. doi: 10.1213/ANE.0000000000003594. PMID 30198928
- [Background] Jiang J, Ma DX, Li B, Wu AS, Xue FS. Videolaryngoscopy versus direct laryngoscopy for nasotracheal intubation: A systematic review and meta-analysis of randomised controlled trials. J Clin Anesth. 2019 Feb;52:6-16. doi: 10.1016/j.jclinane.2018.08.029. Epub 2018 Aug 25. PMID 30153543
- [Background] O'Shea JE, Thio M, Kamlin CO, McGrory L, Wong C, John J, Roberts C, Kuschel C, Davis PG. Videolaryngoscopy to Teach Neonatal Intubation: A Randomized Trial. Pediatrics. 2015 Nov;136(5):912-9. doi: 10.1542/peds.2015-1028. Epub 2015 Oct 19. PMID 26482669
- [Background] Low D, Healy D, Rasburn N. The use of the BERCI DCI Video Laryngoscope for teaching novices direct laryngoscopy and tracheal intubation. Anaesthesia. 2008 Feb;63(2):195-201. doi: 10.1111/j.1365-2044.2007.05323.x. PMID 18211452
- [Background] Herbstreit F, Fassbender P, Haberl H, Kehren C, Peters J. Learning endotracheal intubation using a novel videolaryngoscope improves intubation skills of medical students. Anesth Analg. 2011 Sep;113(3):586-90. doi: 10.1213/ANE.0b013e3182222a66. Epub 2011 Jun 16. PMID 21680859
- [Background] Sun H, Liu M, Lin Z, Jiang H, Niu Y, Wang H, Chen S. Comprehensive identification of 125 multifarious constituents in Shuang-huang-lian powder injection by HPLC-DAD-ESI-IT-TOF-MS. J Pharm Biomed Anal. 2015 Nov 10;115:86-106. doi: 10.1016/j.jpba.2015.06.013. Epub 2015 Jun 30. PMID 26177215
- [Background] Lingappan K, Arnold JL, Fernandes CJ, Pammi M. Videolaryngoscopy versus direct laryngoscopy for tracheal intubation in neonates. Cochrane Database Syst Rev. 2018 Jun 4;6(6):CD009975. doi: 10.1002/14651858.CD009975.pub3. PMID 29862490
- [Background] Goto T, Gibo K, Hagiwara Y, Morita H, Brown DF, Brown CA 3rd, Hasegawa K; Japanese Emergency Medicine Network Investigators. Multiple failed intubation attempts are associated with decreased success rates on the first rescue intubation in the emergency department: a retrospective analysis of multicentre observational data. Scand J Trauma Resusc Emerg Med. 2015 Jan 16;23:5. doi: 10.1186/s13049-014-0085-8. PMID 25700237
- [Background] Goto T, Watase H, Morita H, Nagai H, Brown CA 3rd, Brown DF, Hasegawa K; Japanese Emergency Medicine Network Investigators. Repeated attempts at tracheal intubation by a single intubator associated with decreased success rates in emergency departments: an analysis of a multicentre prospective observational study. Emerg Med J. 2015 Oct;32(10):781-6. doi: 10.1136/emermed-2013-203473. Epub 2014 Dec 31. PMID 25552546
- [Background] Sakles JC, Chiu S, Mosier J, Walker C, Stolz U. The importance of first pass success when performing orotracheal intubation in the emergency department. Acad Emerg Med. 2013 Jan;20(1):71-8. doi: 10.1111/acem.12055. PMID 23574475
- [Background] Mort TC. Emergency tracheal intubation: complications associated with repeated laryngoscopic attempts. Anesth Analg. 2004 Aug;99(2):607-13, table of contents. doi: 10.1213/01.ANE.0000122825.04923.15. PMID 15271750
- [Background] Grunwell JR, Kamat PP, Miksa M, Krishna A, Walson K, Simon D, Krawiec C, Breuer R, Lee JH, Gradidge E, Tarquinio K, Shenoi A, Shults J, Nadkarni V, Nishisaki A; National Emergency Airway Registry for Children (NEAR4KIDS) and the Pediatric Acute Lung Injury and Sepsis (PALISI) Network. Trend and Outcomes of Video Laryngoscope Use Across PICUs. Pediatr Crit Care Med. 2017 Aug;18(8):741-749. doi: 10.1097/PCC.0000000000001175. PMID 28492404
- [Background] Abdelgadir IS, Phillips RS, Singh D, Moncreiff MP, Lumsden JL. Videolaryngoscopy versus direct laryngoscopy for tracheal intubation in children (excluding neonates). Cochrane Database Syst Rev. 2017 May 24;5(5):CD011413. doi: 10.1002/14651858.CD011413.pub2. PMID 28539007
- [Background] Galvez JA, Acquah S, Ahumada L, Cai L, Polanski M, Wu L, Simpao AF, Tan JM, Wasey J, Fiadjoe JE. Hypoxemia, Bradycardia, and Multiple Laryngoscopy Attempts during Anesthetic Induction in Infants: A Single-center, Retrospective Study. Anesthesiology. 2019 Oct;131(4):830-839. doi: 10.1097/ALN.0000000000002847. PMID 31335549
- [Background] Graciano AL, Tamburro R, Thompson AE, Fiadjoe J, Nadkarni VM, Nishisaki A. Incidence and associated factors of difficult tracheal intubations in pediatric ICUs: a report from National Emergency Airway Registry for Children: NEAR4KIDS. Intensive Care Med. 2014 Nov;40(11):1659-69. doi: 10.1007/s00134-014-3407-4. Epub 2014 Aug 27. PMID 25160031
- [Background] Nishisaki A, Turner DA, Brown CA 3rd, Walls RM, Nadkarni VM; National Emergency Airway Registry for Children (NEAR4KIDS); Pediatric Acute Lung Injury and Sepsis Investigators (PALISI) Network. A National Emergency Airway Registry for children: landscape of tracheal intubation in 15 PICUs. Crit Care Med. 2013 Mar;41(3):874-85. doi: 10.1097/CCM.0b013e3182746736. PMID 23328260
- [Background] Garcia-Marcinkiewicz AG, Adams HD, Gurnaney H, Patel V, Jagannathan N, Burjek N, Mensinger JL, Zhang B, Peeples KN, Kovatsis PG, Fiadjoe JE; PeDI Collaborative. A Retrospective Analysis of Neuromuscular Blocking Drug Use and Ventilation Technique on Complications in the Pediatric Difficult Intubation Registry Using Propensity Score Matching. Anesth Analg. 2020 Aug;131(2):469-479. doi: 10.1213/ANE.0000000000004393. PMID 31567318